CLINICAL TRIAL: NCT05116904
Title: Chronobiological Characterization of Smith Magenis Syndrome and Autism Spectrum Disorders in Paediatric Age
Brief Title: Smith Magenis Syndrome and Autism Spectrum Disorders
Acronym: SMS/TSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL20_0682
Record Dates: First submitted 2021-10-21; First posted 2021-11-11 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Smith-Magenis Syndrome; Autism Spectrum Disorder
Keywords: Sleep disorders; Chronobiology; Smith Magenis Syndrome; Paediatrics; Pupillary reflex; Circadian rhythm; Melatonin; Autism Spectrum Disorder
MeSH Terms: conditions — Smith-Magenis Syndrome; Autism Spectrum Disorder; Sleep Wake Disorders | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with Smith Magenis Syndrome (Other)
  Interventions: Other: Assessment
- Children with Autism Spectrum Disorders (Other)
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Pupil reflex and melatonin profile, circadian profile assessment

SUMMARY:
Autism Spectrum Disorders (ASD) are a neurodevelopmental disorder. Their prevalence is estimated at around 0.4% of the general population worldwide. Their early onset and chronic nature make them a disabling disorder, all the more so as there is a high prevalence of sleep disorders in these populations, estimated at between 50 and 80%, with many complaints of insomnia in particular. These sleep disorders may result from biological, psychological, social, environmental and family factors.

Smith Magenis Syndrome (SMS) is a complex disorder characterized by severe neurological, psychological and behavioral disorders including sleep-wake rhythm disorders. It is a rare disease with a prevalence of 1/25 000.

These sleep disorders observed could be the consequence of a general dysregulation of the circadian system, since SMS patients show an inversion of the melatonin secretion profile (with a totally abnormal diurnal peak) and in patients with autism spectrum disorders, an overall reduction in melatonin secretion.

These sleep-wake disturbances cycle could play a significant role in learning deficits and in the frequency and severity of behavioral abnormalities observed in SMS and ASD.

In this project, investigators propose to study the mechanisms involved in the sleep-wake cycle disorders observed in Smith Magenis and Autism Spectrum children, in particular by evaluating the quality of the pupillary reflex using a pupillometer. The pupillary reflex is a simple and non-invasive method to test light sensitivity and the photobiological mechanisms involved.

In this way, investigators want to evaluate the diurnal profile of the pupillary reflex in children with Smith Magenis syndrome and with Autism Spectrum Disorders in relation to the diurnal melatonin profile.

Investigators will complete this study by determining the chronobiological profile of these patients by measuring different variables:

* Diurnal cortisol and amylase profile
* 24h body temperature and heart rate profile
* Urinary cortisol and 6-sulfatoxymelatonin (major metabolite of melatonin) profiles
* Daytime sleepiness profile measured subjectively by questionnaire and objectively via a waking EEG recording.
* Actimetry at home
* Polysomnography
* A neurocognitive and behavioural assessment

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed Smith Magenis syndrome (microdeletion of the short arm of chromosome 17 or mutation of the RAI1 gene; obtained by FISH, CGH-array or molecular biology) and children with neuropsychologically confirmed autism spectrum disorder, with no genetic pathology found.
* Aged 5-12 years
* Consent form signed by the parent(s)
* Requiring a sleep assessment in the Hopital Femme Mère Enfant paediatric sleep unit of Pr Franco
* Affiliation to a social security system.

Exclusion Criteria:

* Associated ophthalmological disorders that do not allow the photomotor reflex to be studied: optic neuritis, glaucoma and retinitis pigmentosa.
* Algic child (risk of measurement bias: when a patient is in pain his pupils dilate and we observe a greater amplitude in the photomotor reflex), defined by a score on the FPS-R Face Scale >4/10.

Only for SMS patients:

- Dyschromatopsia detected in consultation with a rapid Ishihara test adapted to the child's cognitive level, if necessary supplemented by a test performed by ophthalmologists.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Measurement of the percentage change between pupil diameter at the end of light exposure and before exposure | One day
  This measurement will allow to evaluate the diurnal profile of the pupillary reflex and will be measured by a NeuroLight pupillometer (IDMed).
  This measurement will be done every 2 hours from 8am to 8pm, for one day
Measurement of salivary melatonin levels | One day
  This measurement will allow to evaluate the diurnal melatonin profile and will be evaluated using saliva samples.
  This measurement will be done every 2 hours from 8am to 8pm, for one day

SECONDARY OUTCOMES:
Determination of the chronobiological profile : Salivary cortisol levels | Every 2 hours from 8am to 8pm, for one day
  Salivary cortisol levels will be evaluated using saliva samples
Determination of the chronobiological profile : Amylase levels | Every 2 hours from 8am to 8pm, for one day
  Amylase levels will be evaluated using saliva samples
Determination of the chronobiological profile : Urinary 6-sulfatoxymelatonin level | over 24hours
  Urinary 6-sulfatoxymelatonin level will be evaluated using urinary samples
Determination of the chronobiological profile : Urinary cortisol level | over 24hours
  Urinary cortisol level will be evaluated using urinary samples
Determination of the chronobiological profile : Variations in body temperature in degrees | over 24hours
  Body temperature will be measured by ibuttonR placed on the surface of the skin
Determination of the chronobiological profile : Assessment of sleepiness by questionnaire (numerical score) | Every 2 hours from 8am to 8pm, for one day
  The Karolinska questionnaire will be carried out at the time of salivary sampling and pupil diameter measurement and the score obtained will be compared with the salivary melatonin level.
Determination of the chronobiological profile : Assessment of sleepiness by spectral analysis (EEG) | Every 2 hours from 8am to 8pm, for one day
  Somnolence will be evaluated by calculating power spectrum in several frequency bands.
Determination of the chronobiological profile : Sleep assessment by actimetry | 2 weeks
  Home activity monitor during an outpatient recording with a watch in order to assess the sleep wake rhythm at home
Determination of the chronobiological profile :Sleep assessment by Polysomnography | 24 hours
  Polysomnography during hospitalization in order to assess the structure of sleep
Neuropsychological assessment | One day
  WISC +/- Vineland

CONTACTS AND LOCATIONS:
Overall Officials: Patricia FRANCO, PhD, Principal Investigator — Service Épilepsie-Sommeil-Explorations Fonctionnelles Neurologiques Pédiatriques, Hôpital Femme-Mère-Enfant, Hospices Civils de Lyon
Locations (2):
- France (2):
  - Service Épilepsie-Sommeil-Explorations Fonctionnelles Neurologiques Pédiatriques Hôpital Femme-Mère-Enfant HCL, Bron
  - GénoPsy, Reference Center for Diagnosis and Management of Genetic Psychiatric Disorders, Centre Hospitalier le Vinatier and EDR-Psy Q19 Team (Centre National de la Recherche Scientifique & Lyon 1 Claude Bernard University), Bron

IPD SHARING:
Plan to Share IPD: No